CLINICAL TRIAL: NCT03693365
Title: The Reliability of Noninvasive Effective Pulmonary Blood Flow to Detect Fluid Responsiveness During a Positive End-expirator Trial in Ventilated Patients
Brief Title: Fluid Responsiveness Tested by the Effective Pulmonary Blood Flow During a Positive End-expiratory Trial
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 291917072018
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases
Keywords: Carbon dioxide; Pulmonary blood flow; Ventilation
MeSH Terms: conditions — Cardiovascular Diseases; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgeries: Patients undergoing surgery with general anesthesia and controlled mechanical ventilation with indication of invasive arterial blood pressure.
  Classification ASA 2-4
  Interventions: Procedure: PEEP trial

INTERVENTIONS:
Procedure: PEEP trial — Positive end-expiratory pressure (PEEP) is increased from 5 to 10 cmH2O during one minute.

SUMMARY:
Fluid responsiveness is difficult to assess at the bedside. The accuracy of published techniques to detect preload-dependent patients have many pitfalls and limitations. The present study test the role of noninvasive effective pulmonary blood flow measured by expired carbon dioxide to detect fluid responsivess in mechanically ventilated patients.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to test the accuracy of the non-invasive effective pulmonary blood flow measured by the capnodynamic methodology for detect preload-dependent patients.

Fourty patients undergoing mechanical ventilation during surgery will be studied. Preload-depency (fluid responsiveness) will be tested during an increase in end-expiratory pressure (PEEP) from 5 to 10 cmH2O during one minute. Pulse pressure variation will be use as the reference method to detect preload-dependency. The effective pulmonary blood flow will be continuously recorded during the PEEP maneuver. Receiver Operator Curves will be used to detect fluid responsiveness taking a pulse pressure variation higher than 13%.The corresponding cut off value for the effective pulmonary blood flow signal will be determined..

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Programmed cardiac and noncardiac surgeries
* Need of invasive arterial blood pressure monitoring.

Exclusion Criteria:

* Emergency surgeries.
* Acute pulmonary diseases
* Arrhytmias
* Congestive cardiac failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac and noncardiac surgery patients ASA 2-4
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Fluid responsivess assessment with the effective pulmonary blood flow | 10 months
  Comparison between standard method (pulse pressure variation) with a new method of fluid responsiveness (Effective pulmonary blood flow).

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Principal Investigator — Hospital Privado de Comunidad de Mar del Plata
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tusman G, Groisman I, Maidana GA, Scandurra A, Arca JM, Bohm SH, Suarez-Sipmann F. The Sensitivity and Specificity of Pulmonary Carbon Dioxide Elimination for Noninvasive Assessment of Fluid Responsiveness. Anesth Analg. 2016 May;122(5):1404-11. doi: 10.1213/ANE.0000000000001047. PMID 26505574